CLINICAL TRIAL: NCT03096847
Title: A National Phase IIIb, Multi-center, Open Label Study for Women and Men With Hormone-receptor Positive, HER-2 Negative Locally Advanced or Metastatic Breast Cancer Treated With Ribociclib (LEE011) in Combination With Letrozole
Brief Title: Study for Women and Men With Hormone-receptor Positive Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011XDE01; CLEE011XDE01 (Other: Novartis); 2016-002556-24 (EudraCT Number)
Record Dates: First submitted 2017-03-10; First posted 2017-03-30 (Actual); Results first posted 2021-05-19 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Advanced Metastatic Breast Cancer
Keywords: ribociclib; LEE011; RIBECCA; breast cancer; breast carcinoma; HR-positive; HER2-negative; advanced breast cancer; Letrozole; CDK4/6; breast lump; HER2 positive; metastatic breast cancer; breast cancer positive for human epidermal growth factor receptor 2 (HER2) HER2 positive metastatic breast cancer; breast cancer progression; estrogen-receptor (ER) positive(+) breast cancer; Paget's disease
MeSH Terms: conditions — Breast Neoplasms; Osteitis Deformans | interventions — ribociclib; Letrozole; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ribociclib + letrozole cohort A (Experimental): ribociclib + letrozole cohort A - postmenopausal women, or men; naïve.
  All patients received ribociclib 600mg p.o. daily + Letrozole 2.5 mg p.o. daily.
  Interventions: Drug: ribociclib; Drug: letrozole; Drug: goserelin
- ribociclib + letrozole cohort B1 (Experimental): ribociclib + letrozole cohort B1 - premenopausal women or perimenopausal women; naïve
  All patients received ribociclib 600mg p.o. daily + Letrozole 2.5 mg p.o. daily.
  Premenopausal patients additionally received goserelin 3.6 mg i.m. monthly
  Interventions: Drug: ribociclib; Drug: letrozole; Drug: goserelin
- ribociclib + letrozole cohort B2 (Experimental): ribociclib + letrozole cohort B2 - premenopausal women or perimenopausal women or postmenopausal women, or men; pre-treated.
  All patients received ribociclib 600mg p.o. daily + Letrozole 2.5 mg p.o. daily.
  Premenopausal patients additionally received goserelin 3.6 mg i.m. monthly
  Interventions: Drug: ribociclib; Drug: letrozole; Drug: goserelin

INTERVENTIONS:
Drug: ribociclib — All patients with oestrogen receptor positive advanced or metastatic breast cancer were treated with oral ribociclib at a dose of 600mg daily and oral letrozole 2.5mg daily. The study treatment for an individual patient began on Study Day 1 and continued until 80 weeks after the last patient enrolled the study or until disease progression, unacceptable toxicity, death or early discontinuation from the study for any other reason, whichever occured first.
  Other Names: LEE011
Drug: letrozole — All patients with oestrogen receptor positive advanced or metastatic breast cancer were treated with oral ribociclib at a dose of 600mg daily and oral letrozole 2.5mg daily. The study treatment for an individual patient began on Study Day 1 and continued until 80 weeks after the last patient enrolled the study or until disease progression, unacceptable toxicity, death or early discontinuation from the study for any other reason, whichever occured first.
Drug: goserelin — Premenopausal patients additionally received goserelin 3.6mg as monthly implant

SUMMARY:
This was a national, multi-center, open-label, phase IIIb trial to determine the efficacy and safety of treatment with ribociclib (LEE011) plus letrozole in patients with HR+, HER2-negative advanced (recurrent or metastatic) breast cancer. Patients were treated with daily doses of 600 mg ribociclib (3-weeks-on/1-week-off schedule) in combination with 2.5 mg letrozole daily (continuous dosing). Dose adjustments (dose reduction or interruption) according to safety findings were allowed.

DETAILED DESCRIPTION:
The main purpose of this study was to collect additional efficacy and safety data for the combination of ribociclib and letrozole in a patient population broader than the MONALEESA-2 study (NCT01958021 / CLEE011A2301), and to provide access to ribociclib to patients for which available treatment options are unsatisfactory treatment alternatives until the drug is approved for this indication. Furthermore, this trial aimed to collect data for the combination of ribociclib and letrozole in the context of current local routine therapy algorithms for the treatment of metastatic and advanced breast cancer.

This multi-center, open-label, single-arm study aimed to evaluate the efficacy, safety, and quality of life for the combination of ribociclib and letrozole in a patient population than in the MONALEESA-2 study, i.e. in patients pretreated with one line of chemotherapy and/or a maximum of two lines of endocrine therapy as well as premenopausal patients, without limitations regarding the disease free interval after adjuvant therapy.

For ethical reasons no endocrine comparator drugs were investigated in this study. The duration of study treatment of 80 weeks was adequate to determine the primary, secondary and exploratory study parameters. The sample size was suitable to estimate the clinical benefit rate (CBR) in this patient population with reasonable precision.

Goserelin was used in premenopausal patients, since it was shown that ovarian suppression of estrogen release with luteinizing hormone-releasing hormone agonists (LHRHa) (such as goserelin) is effective in preventing relapse in premenopausal women with early stage ER+ breast cancer (Klijn et al. 2001).

The efficacy and safety of ribociclib in combination with letrozole for the treatment of postmenopausal women with advanced or metastatic breast cancer vs. placebo (i.e., letrozole alone) was already demonstrated in the preceding, pivotal MONALESSA-2 study. Thus, for ethical reasons no endocrine comparator drugs were investigated in the present RIBECCA study.

Generally, the single-arm, open-label design and the broadening of the study population (compared to the pivotal MONALESSA-2 study) in the RIBECCA study was deemed appropriate to further evaluate the efficacy and safety of ribociclib plus letrozole among breast cancer patients in a treatment setting closer to routine care. The duration of study treatment of up to 80 weeks was considered adequate to determine the primary, secondary and exploratory study parameters. Moreover, the sample size was suitable to estimate the CBR in this patient population with reasonable precision.

ELIGIBILITY:
Inclusion Criteria:

* Patient is an adult, ≥ 18 years old at the time of informed consent and has signed informed consent before any trial related activities and according to local guidelines
* Women and men with advanced (locoregionally recurrent or metastatic) breast cancer not amenable to curative therapy.
* Patient has a histologically and/or cytologically confirmed diagnosis of estrogen-receptor positive and/or progesterone receptor positive and HER2-negative breast cancer by local laboratory. Local pathology is sufficient for assessment.
* Patient must have either:

  1. Measurable disease, i.e., at least one measurable lesion as per RECIST 1.1 criteria ).
  2. Bone lesions: lytic or mixed (lytic + sclerotic) in the absence of measurable disease
  3. Non-measurable disease
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤2

Exclusion Criteria

* Patient who received any CDK4/6 inhibitor or any mTOR inhibitor.
* Patient has a known hypersensitivity to any of the excipients of ribociclib or letrozole
* Patients with current inflammatory breast cancer.
* Patient has received > 1 chemotherapy for the treatment of advanced/metastatic breast cancer
* Patient has received > 2 endocrine therapies for the treatment of advanced/metastatic breast cancer
* Patient has central nervous system (CNS) involvement. If patient is fulfilling the following 3 criteria she/he is eligible for the trial.

  1. completed prior therapy (including radiation and/or surgery) for CNS metastases ≥ 28 days prior to the start of study and
  2. CNS tumor is clinically stable at the time of screening and
  3. Patient is not receiving steroids and enzyme inducing anti-epileptic medications for brain metastases
* Patient has active cardiac disease or a history of cardiac dysfunction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2020-02-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (67):
- Germany (67):
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Langen, Hesse
  - Novartis Investigative Site, Recklinghausen, North Rhine-Westphalia
  - Novartis Investigative Site, Lübeck, Schleswig-Holstein
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bottrop
  - Novartis Investigative Site, Böblingen
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Esslingen am Neckar
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Fürstenwalde
  - Novartis Investigative Site, Fürth
  - Novartis Investigative Site, Georgsmarienhütte
  - Novartis Investigative Site, Goslar
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Hildesheim
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Kulmbach
  - Novartis Investigative Site, Landshut
  - Novartis Investigative Site, Leer
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, Mönchengladbach
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Neuruppin
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Offenbach
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Passau
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Ravensburg
  - Novartis Investigative Site, Rotenburg (Wümme)
  - Novartis Investigative Site, Saarbrücken
  - Novartis Investigative Site, Schweinfurt
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Suhl
  - Novartis Investigative Site, Torgau
  - Novartis Investigative Site, Trier
  - Novartis Investigative Site, Troisdorf
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Velbert
  - Novartis Investigative Site, Völklingen
  - Novartis Investigative Site, Weinheim
  - Novartis Investigative Site, Wetzlar
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigative Site, Würzburg

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Peuker CA, Yaghobramzi S, Grunert C, Keilholz L, Gjerga E, Hennig S, Schaper S, Na IK, Keller U, Brucker S, Decker T, Fasching P, Fehm T, Janni W, Kummel S, Schneeweiss A, Schuler M, Luftner D, Busse A. Treatment with ribociclib shows favourable immunomodulatory effects in patients with hormone receptor-positive breast cancer-findings from the RIBECCA trial. Eur J Cancer. 2022 Feb;162:45-55. doi: 10.1016/j.ejca.2021.11.025. Epub 2021 Dec 23. PMID 34953442
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=729

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 504 participants were entered into the study, but 2 of these participants were not treated. The full analysis set is comprised of the 504 participants minus 17 participants, whose data were removed because of inspection findings, to equal 487 participants. This full analysis set includes the 2 participants who were entered into the study but were not treated.
  502 participants were treated; these 502 participants are included in the safety set.
Groups:
- Ribociclib + Letrozole Cohort A: postmenopausal women, or men; naïve.
  All patients received ribociclib 600mg p.o. daily + Letrozole 2.5 mg p.o. daily.
- Ribociclib + Letrozole Cohort B1: premenopausal women or perimenopausal women; naïve
  All patients received ribociclib 600mg p.o. daily + Letrozole 2.5 mg p.o. daily.
  Premenopausal patients additionally received goserelin 3.6 mg i.m. monthly
- Ribociclib + Letrozole Cohort B2: premenopausal women or perimenopausal women or postmenopausal women, or men; pre-treated.
  All patients received ribociclib 600mg p.o. daily + Letrozole 2.5 mg p.o. daily.
  Premenopausal patients additionally received goserelin 3.6 mg i.m. monthly
Period: Overall Study
Arm/Group | Ribociclib + Letrozole Cohort A | Ribociclib + Letrozole Cohort B1 | Ribociclib + Letrozole Cohort B2
Started (participants who started treatment) | 319 | 26 | 157
Full Analysis Set | 307 | 26 | 154
Completed (Completed study) | 100 (Only the primary reason for disc. is included in this table.) | 6 (Only the primary reason for disc. is included in this table.) | 19 (Only the primary reason for disc. is included in this table.)
Not Completed | 219 | 20 | 138
Not completed — Other | 2 | 1 | 2
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Death | 6 | 0 | 2
Not completed — Protocol Violation | 3 | 0 | 6
Not completed — Physician Decision | 12 | 2 | 8
Not completed — Withdrawal by Subject | 24 | 1 | 12
Not completed — Adverse Event | 72 | 6 | 28
Not completed — Progressive disease | 97 | 10 | 78
Not completed — Non-compliance with study medication | 1 | 0 | 0
Not completed — New therapy for study indication | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ribociclib + Letrozole Cohort A | Ribociclib + Letrozole Cohort B1 | Ribociclib + Letrozole Cohort B2 | Total
Number analyzed (Participants) | 319 | 26 | 157 | 502
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 143 | 26 | 87 | 256
  >=65 years | 176 | 0 | 70 | 246
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.7 (10.1) | 46.5 (4.9) | 62.8 (12.8) | 63.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 315 | 26 | 156 | 497
  Male | 4 | 0 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 312 | 24 | 151 | 487
  More than one race | 1 | 0 | 3 | 4
  Unknown or Not Reported | 6 | 0 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR) in Women and Men With Hormone Receptor Positiv, HER-2 Negative Breast Cancer Treated With Ribocilib and Letrozole
Description: Clinical Benefit Rate (CBR) after 24 weeks of treatment as defined by RECIST 1.1 as percentage of patients with Complete Response (CR), Partial response (PR) or Stable disease (SD) lasting 24 weeks or longer as well as patients with Non-complete response, nonprogressive disease (NCRNPD).
Time Frame: At 24 weeks after last patient enrolled in trial
Population: Full Analysis Set. Please note that the statistical significance test (test comparing groups) i.e., statistical analysis was not applicable for this outcome measure, since the primary objective was to assess the rate (per cohort) and not to compare two or more treatment arms, as this was a non-randomized, single arm open label trial.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Total: Cohort A and Cohort B combined
Arm/Group | Ribociclib + Letrozole Cohort A | Ribociclib + Letrozole Cohort B1 | Ribociclib + Letrozole Cohort B2 | Total
Number analyzed (Participants) | 307 | 26 | 154 | 487
Percentage of Participants
  CBR by week 24 (= BOR of CR or PR or SD or NCRNPD(Confirmed Best Overall Response (BOR)) | 63.2 [57.5 to 68.6] | 57.7 [36.9 to 76.6] | 56.5 [48.3 to 64.5] | 60.8 [56.3 to 65.1]
  CBR by week 24 (= BOR of CR or PR or SD or NCRNPD (non-confirmed BOR) | 71.7 [66.3 to 76.6] | 69.2 [48.2 to 85.7] | 64.3 [56.2 to 71.8] | 69.2 [64.9 to 73.3]

2. Secondary Outcome: Progression Free Survival (PFS) for Different Populations - Kaplan-Meier Estimates (%, 95% CI)
Description: PFS based on radiologic assessment by investigator using RECIST 1.1 criteria
Time Frame: At week 24 , week 48 and week 72
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ribociclib + Letrozole Cohort A | Ribociclib + Letrozole Cohort B1 | Ribociclib + Letrozole Cohort B2
Number analyzed (Participants) | 307 | 26 | 154
Percentage of Participants
  Kaplan-Meier estimates (%, 95% CI) - Week 24 | 73.1 [67.3 to 77.9] | 67.0 [44.7 to 82.0] | 63.8 [55.2 to 71.3]
  Kaplan-Meier estimates (%, 95% CI) - Week 48 | 61.9 [55.7 to 67.5] | 58.7 [36.8 to 75.2] | 47.5 [38.7 to 55.7]
  Kaplan-Meier estimates (%, 95% CI) - week 72 | 54.5 [48.1 to 60.5] | 49.6 [28.6 to 67.6] | 39.3 [30.8 to 47.6]

3. Secondary Outcome: Progression Free Survival (PFS) for Different Populations - Median Time to Progression or Death With 95% CI [Months]
Description: PFS based on radiologic assessment by investigator using RECIST 1.1 criteria
Time Frame: Up to approximately month 25
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ribociclib + Letrozole Cohort A | Ribociclib + Letrozole Cohort B1 | Ribociclib + Letrozole Cohort B2
Number analyzed (Participants) | 307 | 26 | 154
Months | 21.8 [13.9 to 25.3] | 16.5 [3.2 to NA] — The upper limit was not estimable. Existence of the confidence limits does not directly depend on the Kaplan-Meier curve itself (dropping below 0.75, 0.5 or 0.25), but on the curves that represent the confidence limits (CL) for the survivor function. They envelop the Kaplan-Meier curve. | 8.8 [8.1 to 16.3]

4. Secondary Outcome: Overall Survival (OS) - Kaplan-Meier Estimates (%, 95% CI)
Description: Overall survival (OS) defined as the time from date of start of treatment to date of death due to any cause. For the Kaplan-Meier estimates (%, 95% CI), the probability of survival at week 24, 48 and 72 is reported below.
Time Frame: At Week 24, Week 48 and Week 72
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ribociclib + Letrozole Cohort A | Ribociclib + Letrozole Cohort B1 | Ribociclib + Letrozole Cohort B2
Number analyzed (Participants) | 307 | 26 | 154
Percentage of Participants
  Kaplan-Meier estimates (%, 95% CI) - Week 24 | 98.6 [96.4 to 99.5] | 100.0 [100.0 to 100.0] | 93.9 [88.5 to 96.8]
  Kaplan-Meier estimates (%, 95% CI) - Week 48 | 93.3 [89.7 to 95.7] | 87.5 [66.1 to 95.8] | 86.1 [79.2 to 90.8]
  Kaplan-Meier estimates (%, 95% CI) - Week 72 | 89.7 [85.5 to 92.7] | 87.5 [66.1 to 95.8] | 81.0 [73.5 to 86.6]

5. Secondary Outcome: Overall Survival (OS) - Median Time to Progression or Death With 95% CI [Months]
Description: Overall survival (OS) defined as the time from date of start of treatment to date of death due to any cause.
Time Frame: Up to approximatley 38 months
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ribociclib + Letrozole Cohort A | Ribociclib + Letrozole Cohort B1 | Ribociclib + Letrozole Cohort B2
Number analyzed (Participants) | 307 | 26 | 154
Months | NA [NA to NA] — Not estimable. Existence of the confidence limits does not directly depend on the Kaplan-Meier curve itself (dropping below 0.75, 0.5 or 0.25), but on the curves that represent the confidence limits (CL) for the survivor function. They envelop the Kaplan-Meier curve. | NA [30.9 to NA] — Not estimable. Existence of the confidence limits does not directly depend on the Kaplan-Meier curve itself (dropping below 0.75, 0.5 or 0.25), but on the curves that represent the confidence limits (CL) for the survivor function. They envelop the Kaplan-Meier curve. | NA [31.0 to NA] — Not estimable. Existence of the confidence limits does not directly depend on the Kaplan-Meier curve itself (dropping below 0.75, 0.5 or 0.25), but on the curves that represent the confidence limits (CL) for the survivor function. They envelop the Kaplan-Meier curve.

6. Secondary Outcome: Overall Survival (OS) - Number of Censored Participants and Number of Deaths
Description: Overall survival (OS) defined as the time from date of start of treatment to date of death due to any cause.
Time Frame: Up to approximatley 38 months
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Ribociclib + Letrozole Cohort A | Ribociclib + Letrozole Cohort B1 | Ribociclib + Letrozole Cohort B2
Number analyzed (Participants) | 307 | 26 | 154
Participants
  No. of censored (no death), n | 240 | 17 | 94
  No. of events (deaths due to any cause), n | 67 | 9 | 60

7. Secondary Outcome: Overall Response Rate (ORR) - Kaplan-Meier Estimates (%, 95% CI)
Description: Overall response rate (ORR) is the best overall response (BOR) of complete response (CR) or partial response (PR) as defined by RECIST 1.1.
Time Frame: At week 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ribociclib + Letrozole Cohort A | Ribociclib + Letrozole Cohort B1 | Ribociclib + Letrozole Cohort B2
Number analyzed (Participants) | 307 | 26 | 154
Percentage of Participants
  ORR by week 24 - (BOR of CR or PR) (confirmed) | 22.8 [18.2 to 27.9] | 23.1 [9.0 to 43.6] | 11.7 [7.1 to 17.8]
  ORR by week 24 - (BOR of CR or PR) (unconfirmed) | 24.8 [20.0 to 30.0] | 30.8 [14.3 to 51.8] | 16.2 [10.8 to 23.0]

8. Secondary Outcome: Change From Baseline at Week 24 of Patient Reported Quality of Life (QoL) Via EORTC QLQ-C30
Description: The QLQ-C30 is the core questionnaire of the EORTC QLQ, which has been developed for the assessment of the health-related QOL of cancer patients participating in international clinical trials. Using a linear transformation to standardize the raw scores, all scores finally range from 0 to 100, where a higher score represents a higher response level, e.g., a higher ("better") level of functioning (applies to the first 6 items, items 1 to 6), but a higher ("worse") level of symptoms (applies to the last 9 items, items 7 to 15). There is no aggregated total score, i.e., all scale scores were analyzed separately.
Time Frame: Change from Baseline to Week 24
Population: Full Analysis Set. Included in the analysis are all patients with valid assessment at baseline and week 24. Some questions were conditional branching and thus did not apply to some participants. Also, some participants chose not to answer some questions / items; the responses were accepted as provided by the participants. Also, some participants discontinued during the course of the trial, and thus less measurements were taken at week 24 than at baseline.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Ribociclib + Letrozole Cohort B: premenopausal women or perimenopausal women or postmenopausal women, or men; naïve + pre-treated
  All patients received ribociclib 600mg p.o. daily + Letrozole 2.5 mg p.o.daily.
  Premenopausal patients additionally received goserelin 3.6 mg i.m. monthly
Arm/Group | Ribociclib + Letrozole Cohort A | Ribociclib + Letrozole Cohort B1 | Ribociclib + Letrozole Cohort B2 | Ribociclib + Letrozole Cohort B
Number analyzed (Participants) | 307 | 26 | 154 | 180
Scores on a scale
  Global health status - Change from baseline to Week 24 (C7D1): number analyzed (Participants) | 181 | 15 | 75 | 90
  Global health status - Change from baseline to Week 24 (C7D1) | 8.8 (23.7) | 11.7 (20.8) | 5.0 (26.2) | 6.1 (25.4)
  Physical Functioning - Change from baseline to Week 24 (C7D1): number analyzed (Participants) | 183 | 15 | 75 | 90
  Physical Functioning - Change from baseline to Week 24 (C7D1) | -3.1 (19.9) | -3.6 (10.7) | -2.2 (17.7) | -2.4 (16.7)
  Role Functioning - Change from baseline to Week 24 (C7D1): number analyzed (Participants) | 182 | 15 | 75 | 90
  Role Functioning - Change from baseline to Week 24 (C7D1) | -6.6 (31.9) | -17 (21.8) | -1.3 (34.7) | -3.9 (33.3)
  Emotional Functioning - Change from baseline to Week 24 (C7D1): number analyzed (Participants) | 182 | 15 | 75 | 90
  Emotional Functioning - Change from baseline to Week 24 (C7D1) | -9.6 (24.2) | -9.4 (25.0) | -3.6 (21.8) | -4.6 (22.4)
  Cognitive Functioning - Change from baseline to Week 24 (C7D1): number analyzed (Participants) | 182 | 15 | 75 | 90
  Cognitive Functioning - Change from baseline to Week 24 (C7D1) | 2.7 (23.7) | 2.2 (28.1) | 1.1 (21.6) | 1.3 (22.7)
  Social Functioning - Change from baseline to Week 24 (C7D1): number analyzed (Participants) | 181 | 15 | 75 | 90
  Social Functioning - Change from baseline to Week 24 (C7D1) | -6.9 (27.9) | -16 (21.3) | -5.3 (31.3) | -7.0 (30.0)
  Fatigue - Change from baseline to Week 24 (C7D1): number analyzed (Participants) | 182 | 15 | 75 | 90
  Fatigue - Change from baseline to Week 24 (C7D1) | 6.3 (25.9) | 11.1 (20.6) | 3.9 (27.1) | 5.1 (26.1)
  Nausea / Vomiting - Change from baseline to Week 24 (C7D1): number analyzed (Participants) | 182 | 15 | 75 | 90
  Nausea / Vomiting - Change from baseline to Week 24 (C7D1) | 0.1 (16.7) | 1.1 (22.2) | -4.9 (19.1) | -3.9 (19.7)
  Pain - Change from baseline to Week 24 (C7D1): number analyzed (Participants) | 182 | 15 | 74 | 89
  Pain - Change from baseline to Week 24 (C7D1) | 13.2 (31.9) | 15.6 (24.8) | 9.0 (27.6) | 10.1 (27.1)
  Dyspnoea - Change from baseline to Week 24 (C7D1): number analyzed (Participants) | 182 | 15 | 75 | 90
  Dyspnoea - Change from baseline to Week 24 (C7D1) | 3.8 (32.4) | 4.4 (21.3) | -5.3 (30.5) | -3.7 (29.3)
  Insomnia - Change from baseline to Week 24 (C7D1): number analyzed (Participants) | 183 | 15 | 75 | 90
  Insomnia - Change from baseline to Week 24 (C7D1) | 4.2 (33.2) | 6.7 (31.4) | 4.9 (32.7) | 5.2 (32.3)
  Appetite loss - Change from baseline to Week 24 (C7D1): number analyzed (Participants) | 181 | 15 | 74 | 89
  Appetite loss - Change from baseline to Week 24 (C7D1) | 11.2 (33.7) | 6.7 (28.7) | 1.4 (30.9) | 2.2 (30.5)
  Constipation - Change from baseline to Week 24 (C7D1): number analyzed (Participants) | 183 | 15 | 74 | 89
  Constipation - Change from baseline to Week 24 (C7D1) | -2.7 (26.6) | 2.2 (26.6) | -3.6 (27.9) | -2.6 (27.6)
  Diarrhea - Change from baseline to Week 24 (C7D1): number analyzed (Participants) | 182 | 15 | 74 | 89
  Diarrhea - Change from baseline to Week 24 (C7D1) | 2.6 (24.6) | 0.0 (45.4) | 2.3 (27.2) | 1.9 (30.7)
  Financial Problems - Change from baseline to Week 24 (C7D1): number analyzed (Participants) | 179 | 15 | 73 | 88
  Financial Problems - Change from baseline to Week 24 (C7D1) | 0.2 (27.7) | -4.4 (24.8) | -1.4 (25.1) | -1.9 (24.9)

9. Secondary Outcome: Patient Reported Quality of Life (QoL) Via EORTC BR-23 - Change From Baseline at Week 24 (Cycle 7)
Description: To evaluate health related quality of life (QoL) via EORTC BR-23. The scoring approach for the QLQ-BR23 is identical in principle to that for the function and symptom scales / single items of the QLQ-C30, i.e., all scores finally range from 0 to 100, where a higher score represents a higher response level, e.g., a higher ("better") level of functioning, (applies to the first 4 items, items 1 to 4) but a higher ("worse") level of symptoms (applies to the last 4 items, items 5 to 8).
Time Frame: Baseline and Week 24 (Cycle 7)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ribociclib + Letrozole Cohort A | Ribociclib + Letrozole Cohort B1 | Ribociclib + Letrozole Cohort B2 | Ribociclib + Letrozole Cohort B
Number analyzed (Participants) | 307 | 26 | 154 | 180
Scores on a scale
  EORTC QLQ-BR23 BODY IMAGE during the study - change from baseline at cycle 7: number analyzed (Participants) | 167 | 15 | 72 | 87
  EORTC QLQ-BR23 BODY IMAGE during the study - change from baseline at cycle 7 | -1.5 (18.2) | -0.6 (22.2) | 0.4 (22.7) | 0.2 (22.5)
  EORTC QLQ-BR23 SEXUAL FUNCTIONING during the study - change from baseline at cycle 7: number analyzed (Participants) | 120 | 13 | 60 | 73
  EORTC QLQ-BR23 SEXUAL FUNCTIONING during the study - change from baseline at cycle 7 | -1.1 (17.7) | 0.0 (24.5) | 0.8 (18.0) | 0.7 (19.1)
  EORTC QLQ-BR23 SEXUAL ENJOYMENT during the study - change from baseline at cycle 7: number analyzed (Participants) | 18 | 2 | 18 | 20
  EORTC QLQ-BR23 SEXUAL ENJOYMENT during the study - change from baseline at cycle 7 | -1.9 (31.3) | -17 (23.6) | 7.4 (26.9) | 5.0 (27.1)
  EORTC QLQ-BR23 FUTURE PERSPECTIVE during the study - change from baseline at cycle 7: number analyzed (Participants) | 172 | 15 | 74 | 89
  EORTC QLQ-BR23 FUTURE PERSPECTIVE during the study - change from baseline at cycle 7 | -20 (33.4) | -24 (26.6) | -12 (26.2) | -14 (26.5)
  EORTC QLQ-BR23 SYSTEMATIC THERAPY during the study - change from baseline at cycle 7: number analyzed (Participants) | 180 | 15 | 74 | 89
  EORTC QLQ-BR23 SYSTEMATIC THERAPY during the study - change from baseline at cycle 7 | -9.4 (16.6) | -13 (22.3) | -6.0 (14.9) | -7.1 (16.4)
  EORTC QLQ-BR23 BREAST SYMPTOMS during the study - change from baseline at cycle 7: number analyzed (Participants) | 172 | 15 | 73 | 88
  EORTC QLQ-BR23 BREAST SYMPTOMS during the study - change from baseline at cycle 7 | 3.3 (15.7) | 8.3 (22.7) | 0.9 (17.5) | 2.2 (18.6)
  EORTC QLQ-BR23 ARM SYMPTOMS during the study - change from baseline at cycle 7: number analyzed (Participants) | 175 | 15 | 74 | 89
  EORTC QLQ-BR23 ARM SYMPTOMS during the study - change from baseline at cycle 7 | 4.1 (21.1) | -1.5 (22.6) | -2.1 (18.1) | -2.0 (18.8)
  EORTC QLQ-BR23 HAIR LOSS during the study - change from baseline at cycle 7: number analyzed (Participants) | 23 | 2 | 14 | 16
  EORTC QLQ-BR23 HAIR LOSS during the study - change from baseline at cycle 7 | -22 (43.4) | -17 (23.6) | -14 (33.9) | -15 (32.1)

10. Secondary Outcome: Time to 10% Deterioration in EORTC Global Health Status
Description: Time to 10% deterioration in the European Organisation for Research and Treatment of Cancer (EORTC) global health status
Time Frame: up to approximately 10 months
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Total: Cohorts A, B1 and B2 combined
Arm/Group | Ribociclib + Letrozole Cohort A | Ribociclib + Letrozole Cohort B1 | Ribociclib + Letrozole Cohort B2 | Total
Number analyzed (Participants) | 307 | 26 | 154 | 487
months | 3.3 [2.8 to 4.6] | 3.7 [1.8 to 10.1] | 2.8 [1.8 to 4.6] | 3.0 [2.8 to 4.6]

11. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE)
Description: Adverse Events (AEs) were separated into TEAEs (defined as AEs occurring/worsening from first study drug treatment until 30 days after the last study drug treatment) and AEs in the pre-/post-treatment period.
Time Frame: Up to Week 72
Population: Safety Set
Measure: Number; unit: Number of Participants
Arm/Group | Ribociclib + Letrozole Cohort A | Ribociclib + Letrozole Cohort B1 | Ribociclib + Letrozole Cohort B2
Number analyzed (Participants) | 319 | 26 | 157
Number of Participants
  Total AEs (i.e., Includes any type of AE.) | 318 | 25 | 157
  Serious AEs | 97 | 5 | 45
  Non-serious AEs | 317 | 25 | 157
  AEs with suspected relationship to ribociclib | 302 | 25 | 144
  AEs leading to discontinuation of ribociclib | 76 | 7 | 38
  AEs with fatal outcome | 6 | 0 | 6

12. Post Hoc Outcome: All Collected Deaths
Description: On treatment deaths were collected from FPFT up to 30 days after study drug discontinuation, for a maximum duration of 1150 days (approx 3.15 years). (Treatment duration ranged from 2 days to 1120 days). Deaths post treatment survival follow up were collected after the on- treatment period, up to approx. 3.15 years. Patients who didn't die during the on-treatment period and had not stopped study participation at the time of data cut-off (end of study) were censored.
Time Frame: on-treatment deaths: up to approx 3.15 years; all deaths: approx 3.15 years
Population: Clinical database population - all treated participants
Measure: Number; unit: Participants
Groups:
- Ribociclib + Letrozole Cohort B2: premenopausal women or perimenopausal women or postmenopausal women, or men; pre-treated. All patients received ribociclib 600mg p.o. daily + Letrozole 2.5 mg p.o. daily. Premenopausal patients additionally rec
Arm/Group | Ribociclib + Letrozole Cohort A | Ribociclib + Letrozole Cohort B1 | Ribociclib + Letrozole Cohort B2 | Total
Number analyzed (Participants) | 319 | 26 | 157 | 502
Participants
  on-treatment deaths | 6 | 0 | 6 | 12
  Total deaths: number analyzed (Participants) | 307 | 26 | 154 | 487
  Total deaths | 67 | 9 | 60 | 136

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days, up to a maximum duration of 1150 days (approx. 3.15 years).(Treatment duration ranged from 2 days to 1120 days.)
Description: For this study, disease progression was NOT classified as an Adverse Event.
Groups:
- Total: Total
Arm/Group | Ribociclib + Letrozole Cohort A | Ribociclib + Letrozole Cohort B | Ribociclib + Letrozole Cohort B1 | Ribociclib + Letrozole Cohort B2 | Total
All-Cause Mortality (participants affected / at risk) | 6/319 | 6/183 | 0/26 | 6/157 | 12/502
Serious Adverse Events (participants affected / at risk) | 97/319 | 50/183 | 5/26 | 45/157 | 147/502
Other Adverse Events (participants affected / at risk) | 315/319 | 181/183 | 25/26 | 156/157 | 496/502
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ribociclib + Letrozole Cohort A (N=319) | Ribociclib + Letrozole Cohort B (N=183) | Ribociclib + Letrozole Cohort B1 (N=26) | Ribociclib + Letrozole Cohort B2 (N=157) | Total (N=502)
ANAEMIA (Blood and lymphatic system disorders) | 4 | 4 | 0 | 4 | 8
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 3 | 1 | 2 | 3
HYPERFIBRINOLYSIS (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 2
NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 2 | 0 | 2 | 4
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0 | 3
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 2 | 0 | 2 | 4
BRADYARRHYTHMIA (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
CARDIAC FAILURE (Cardiac disorders) | 1 | 1 | 0 | 1 | 2
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
HYPERTHYROIDISM (Endocrine disorders) | 1 | 0 | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 2
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
CONSTIPATION (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 2
DIARRHOEA (Gastrointestinal disorders) | 3 | 1 | 0 | 1 | 4
GASTRITIS (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 3
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
ILEUS (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 2
INTESTINAL STRANGULATION (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
NAUSEA (Gastrointestinal disorders) | 7 | 2 | 0 | 2 | 9
VOMITING (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 3
CHEST PAIN (General disorders) | 1 | 1 | 0 | 1 | 2
COMPLICATION OF DEVICE INSERTION (General disorders) | 0 | 1 | 0 | 1 | 1
DEATH (General disorders) | 1 | 0 | 0 | 0 | 1
FATIGUE (General disorders) | 0 | 2 | 0 | 2 | 2
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 2 | 5 | 0 | 5 | 7
IMPAIRED HEALING (General disorders) | 1 | 2 | 0 | 2 | 3
OEDEMA PERIPHERAL (General disorders) | 1 | 0 | 0 | 0 | 1
PAIN (General disorders) | 1 | 1 | 0 | 1 | 2
PYREXIA (General disorders) | 6 | 1 | 0 | 1 | 7
BILE DUCT STENOSIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
BILIARY COLIC (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 2
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 5 | 1 | 0 | 1 | 6
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 1
HEPATOTOXICITY (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
JAUNDICE (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
ABDOMINAL ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 1
ABSCESS JAW (Infections and infestations) | 0 | 1 | 0 | 1 | 1
APPENDICITIS (Infections and infestations) | 0 | 1 | 0 | 1 | 1
ATYPICAL PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 0 | 1
BRONCHITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 1
CHOLECYSTITIS INFECTIVE (Infections and infestations) | 1 | 0 | 0 | 0 | 1
CYSTITIS (Infections and infestations) | 0 | 1 | 0 | 1 | 1
CYSTITIS ESCHERICHIA (Infections and infestations) | 0 | 1 | 0 | 1 | 1
DEVICE RELATED INFECTION (Infections and infestations) | 0 | 2 | 0 | 2 | 2
DIVERTICULITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 1
EMPHYSEMATOUS CHOLECYSTITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 1
ERYSIPELAS (Infections and infestations) | 3 | 0 | 0 | 0 | 3
ESCHERICHIA INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 1
FEBRILE INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 1
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 | 1 | 0 | 1 | 2
HELICOBACTER GASTRITIS (Infections and infestations) | 0 | 1 | 0 | 1 | 1
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 1 | 0 | 0 | 0 | 1
INFLUENZA (Infections and infestations) | 0 | 1 | 0 | 1 | 1
MASTITIS (Infections and infestations) | 0 | 1 | 0 | 1 | 1
PNEUMONIA (Infections and infestations) | 8 | 2 | 0 | 2 | 10
PROTEUS INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 1
PYELONEPHRITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 1
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 1
SEPSIS (Infections and infestations) | 1 | 1 | 0 | 1 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 3 | 0 | 0 | 0 | 3
UROSEPSIS (Infections and infestations) | 2 | 0 | 0 | 0 | 2
ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
FALL (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 3
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1
JAW FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
POSTOPERATIVE ADHESION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 3
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 5 | 1 | 0 | 1 | 6
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 1 | 0 | 1 | 4
BLOOD BILIRUBIN INCREASED (Investigations) | 1 | 1 | 0 | 1 | 2
C-REACTIVE PROTEIN INCREASED (Investigations) | 1 | 0 | 0 | 0 | 1
HAEMOGLOBIN DECREASED (Investigations) | 1 | 0 | 0 | 0 | 1
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 1 | 1 | 0 | 1
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 1 | 1 | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 2
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
HYPOPHAGIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 2
BONE LESION (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 2 | 4
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
MOBILITY DECREASED (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 2
OSTEITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 2
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 1
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 2
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 1
METASTASES TO SPINE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 1
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
SQUAMOUS CELL CARCINOMA OF THE TONGUE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 1
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 1
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2 | 0 | 0 | 0 | 2
DIZZINESS (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
HEADACHE (Nervous system disorders) | 0 | 1 | 0 | 1 | 1
MONOPLEGIA (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
PARAESTHESIA (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
PERIPHERAL NERVE LESION (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
SYNCOPE (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
DEVICE LOOSENING (Product Issues) | 0 | 1 | 0 | 1 | 1
DEPRESSION (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1
PANIC ATTACK (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1
SOMATIC SYMPTOM DISORDER (Psychiatric disorders) | 2 | 0 | 0 | 0 | 2
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 5 | 1 | 1 | 0 | 6
HAEMATURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
KIDNEY CONGESTION (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
RENAL DISORDER (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 2
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 2
URETERIC STENOSIS (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
URETEROLITHIASIS (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
URINARY RETENTION (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
PELVIC PAIN (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | 0 | 3 | 12
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
HYPERVENTILATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 3 | 6
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 0 | 1 | 8
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1
CIRCULATORY COLLAPSE (Vascular disorders) | 0 | 1 | 0 | 1 | 1
HYPERTENSION (Vascular disorders) | 0 | 1 | 0 | 1 | 1
HYPERTENSIVE CRISIS (Vascular disorders) | 1 | 0 | 0 | 0 | 1
HYPOTENSION (Vascular disorders) | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ribociclib + Letrozole Cohort A (N=319) | Ribociclib + Letrozole Cohort B (N=183) | Ribociclib + Letrozole Cohort B1 (N=26) | Ribociclib + Letrozole Cohort B2 (N=157) | Total (N=502)
ANAEMIA (Blood and lymphatic system disorders) | 46 | 36 | 7 | 29 | 82
LEUKOPENIA (Blood and lymphatic system disorders) | 76 | 39 | 8 | 31 | 115
LYMPHOPENIA (Blood and lymphatic system disorders) | 7 | 2 | 2 | 0 | 9
NEUTROPENIA (Blood and lymphatic system disorders) | 162 | 88 | 15 | 73 | 250
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 26 | 18 | 1 | 17 | 44
VERTIGO (Ear and labyrinth disorders) | 33 | 17 | 4 | 13 | 50
DRY EYE (Eye disorders) | 23 | 10 | 2 | 8 | 33
LACRIMATION INCREASED (Eye disorders) | 34 | 11 | 2 | 9 | 45
ABDOMINAL PAIN (Gastrointestinal disorders) | 15 | 14 | 5 | 9 | 29
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 33 | 13 | 3 | 10 | 46
CONSTIPATION (Gastrointestinal disorders) | 62 | 32 | 4 | 28 | 94
DIARRHOEA (Gastrointestinal disorders) | 85 | 40 | 8 | 32 | 125
DRY MOUTH (Gastrointestinal disorders) | 28 | 10 | 1 | 9 | 38
DYSPEPSIA (Gastrointestinal disorders) | 25 | 14 | 2 | 12 | 39
NAUSEA (Gastrointestinal disorders) | 130 | 77 | 9 | 68 | 207
STOMATITIS (Gastrointestinal disorders) | 33 | 27 | 4 | 23 | 60
TOOTHACHE (Gastrointestinal disorders) | 9 | 4 | 2 | 2 | 13
VOMITING (Gastrointestinal disorders) | 66 | 31 | 5 | 26 | 97
FATIGUE (General disorders) | 123 | 74 | 15 | 59 | 197
OEDEMA PERIPHERAL (General disorders) | 35 | 22 | 5 | 17 | 57
PYREXIA (General disorders) | 23 | 14 | 4 | 10 | 37
SEASONAL ALLERGY (Immune system disorders) | 4 | 6 | 3 | 3 | 10
BRONCHITIS (Infections and infestations) | 19 | 5 | 1 | 4 | 24
CYSTITIS (Infections and infestations) | 21 | 9 | 3 | 6 | 30
GASTROINTESTINAL INFECTION (Infections and infestations) | 2 | 3 | 2 | 1 | 5
NASOPHARYNGITIS (Infections and infestations) | 94 | 49 | 10 | 39 | 143
URINARY TRACT INFECTION (Infections and infestations) | 31 | 17 | 1 | 16 | 48
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 3 | 3 | 2 | 1 | 6
ARTHROPOD STING (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0 | 2
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 75 | 36 | 6 | 30 | 111
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 66 | 36 | 5 | 31 | 102
BLOOD BILIRUBIN INCREASED (Investigations) | 16 | 1 | 0 | 1 | 17
BLOOD CREATININE INCREASED (Investigations) | 27 | 12 | 2 | 10 | 39
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 17 | 3 | 1 | 2 | 20
BLOOD THYROID STIMULATING HORMONE INCREASED (Investigations) | 0 | 2 | 2 | 0 | 2
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 23 | 14 | 1 | 13 | 37
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 33 | 18 | 5 | 13 | 51
NEUTROPHIL COUNT DECREASED (Investigations) | 40 | 25 | 2 | 23 | 65
WEIGHT DECREASED (Investigations) | 16 | 9 | 0 | 9 | 25
WEIGHT INCREASED (Investigations) | 7 | 4 | 2 | 2 | 11
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 27 | 18 | 2 | 16 | 45
DECREASED APPETITE (Metabolism and nutrition disorders) | 44 | 19 | 1 | 18 | 63
HYPERKALAEMIA (Metabolism and nutrition disorders) | 6 | 4 | 2 | 2 | 10
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 8 | 5 | 2 | 3 | 13
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 57 | 39 | 9 | 30 | 96
BACK PAIN (Musculoskeletal and connective tissue disorders) | 37 | 24 | 4 | 20 | 61
BONE PAIN (Musculoskeletal and connective tissue disorders) | 35 | 15 | 6 | 9 | 50
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 12 | 6 | 2 | 4 | 18
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 21 | 14 | 2 | 12 | 35
MYALGIA (Musculoskeletal and connective tissue disorders) | 18 | 6 | 0 | 6 | 24
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 52 | 23 | 3 | 20 | 75
DIZZINESS (Nervous system disorders) | 26 | 12 | 4 | 8 | 38
DYSGEUSIA (Nervous system disorders) | 20 | 11 | 4 | 7 | 31
HEADACHE (Nervous system disorders) | 56 | 36 | 10 | 26 | 92
HYPOAESTHESIA (Nervous system disorders) | 3 | 5 | 3 | 2 | 8
POLYNEUROPATHY (Nervous system disorders) | 16 | 5 | 1 | 4 | 21
DEPRESSION (Psychiatric disorders) | 7 | 8 | 2 | 6 | 15
INSOMNIA (Psychiatric disorders) | 31 | 26 | 4 | 22 | 57
SLEEP DISORDER (Psychiatric disorders) | 13 | 10 | 4 | 6 | 23
VULVOVAGINAL DRYNESS (Reproductive system and breast disorders) | 4 | 3 | 3 | 0 | 7
COUGH (Respiratory, thoracic and mediastinal disorders) | 53 | 22 | 6 | 16 | 75
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 49 | 25 | 4 | 21 | 74
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 11 | 7 | 5 | 2 | 18
ALOPECIA (Skin and subcutaneous tissue disorders) | 119 | 57 | 5 | 52 | 176
DRY SKIN (Skin and subcutaneous tissue disorders) | 24 | 15 | 3 | 12 | 39
ERYTHEMA (Skin and subcutaneous tissue disorders) | 9 | 10 | 1 | 9 | 19
PRURITUS (Skin and subcutaneous tissue disorders) | 45 | 18 | 3 | 15 | 63
RASH (Skin and subcutaneous tissue disorders) | 47 | 19 | 2 | 17 | 66
HOT FLUSH (Vascular disorders) | 44 | 30 | 11 | 19 | 74
HYPERTENSION (Vascular disorders) | 36 | 11 | 4 | 7 | 47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/47/NCT03096847/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT03096847/SAP_001.pdf